CLINICAL TRIAL: NCT01884389
Title: Randomized Trial of an HIV Navigation Program for Early Palliative Care
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Jacquelyn Slomka, Assistant Professor, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RES121956; R01NR014059 (NIH)
Record Dates: First submitted 2013-06-14; First posted 2013-06-24 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: HIV; Chronic Disease
Keywords: HIV; Chronic disease; Early palliative care; Patient navigation
MeSH Terms: conditions — Chronic Disease | interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patient Navigation (Experimental): Patients are "admitted" to the navigation program, provided through a local community partner agency. Each of these subjects will be assigned an advanced practice nurse (APN) and licensed social worker (LSW) as co-case managers, with their relative contributions depending on the nature of the subject's needs. Level of need (1, 2 or 3) will be confirmed for each patient, and the level will inform the amount of in-person and phone call contacts made to provide on-going support and monitoring of patients. Additionally, this group will meet with the research team for data collection at enrollment and at four 9-month intervals for a total of 5 time points.
  Interventions: Other: Patient Navigation
- Usual Care (No Intervention): The control group will receive "usual care" - medical care and support provided by their primary care provider. They will not receive any of the navigation program services. To provide control for the effects of attention, we will contact these subjects at baseline and every other month thereafter by phone. During these contacts, we will ask a scripted "social" query (e.g. "How are things going for you?"). A subject who raises any health issues or need for specific information will be referred to the primary care provider. Additionally, this group will meet with the research team for data collection at enrollment and at four 9-month intervals for a total of 5 time points.

INTERVENTIONS:
Other: Patient Navigation — Home-based medical and social support services, as an extension of and collaboration with primary care services provided. Phone calls and visits scheduled based on patient's level of need. Communication with primary care team via navigation plan faxed / emailed as needed. Volunteers will also be matched with intervention patients to provide additional support services by phone / in-person visits.
  Arms: Patient Navigation

SUMMARY:
This study is testing a navigation program for early palliative care provided in tandem with HIV primary care for persons living with HIV (PLWH) who are at high risk or mortality and morbidity related to their co-morbid chronic conditions. Participants are enrolled for a period of 36 months, with data collection at enrollment and every 9 months after, for a total of 5 data collection time points. Study participants enrolled will be randomized into one of two groups: control or intervention. Control group participants will receive control calls in between survey data collection time points. Intervention group participants will participate in a Navigation Program which includes home visits and phone calls with an advanced practice nurse (APN) and licensed social worker (LSW), as well as visits / calls by a volunteer if desired. The frequency of visits / calls will be determined based on level of need (high, medium or low).

The specific aims of the study are to: 1) identify needs and preferences for palliative care and advance care planning for PLWH, in order to tailor an existing Navigation Program for this study; 2) test the effectiveness of an HIV Navigation Program intervention on outcomes of quality of life, symptom burden, coping ability, and advance care planning; and 3) determine if effectiveness of the HIV Navigation Program intervention differs by age, gender, ethnicity, education, income level, and level of palliative care service need.

DETAILED DESCRIPTION:
With the advent of effective antiretroviral treatment for HIV has come a marked increase in the number of persons living with HIV/AIDS (PLWHA), with the highest prevalence since the epidemic began of more than 1.2 million. While PLWHA survive longer, they also experience increased burdens of chronic conditions related to lifestyle factors, treatment side effects, and age. PLWHA are a population at great risk for high symptom burden, impaired coping and social functioning, decreased quality of life, and inadequate end-of-life care. The remarkable shift in attitudes towards HIV, from an inevitably fatal disease to a chronic condition, has been accompanied by a lessening emphasis on symptom management and end-of-life planning. However, while mortality from AIDS-defining conditions has decreased, PLWHA continue to have unaddressed needs for coordinated care, symptom management and proactive advance care planning. Palliative care, focused on comprehensive management of physical, psychological, social, and spiritual needs of persons with incurable, progressive illnesses, is a health service uniquely designed to meet these needs. This research project will test a model of early palliative care for PLWHA at high risk of mortality and morbidity. First, focus group methods will be used to explore views of PLWHA regarding their needs for symptom management and social support, and attitudes towards advance care planning and end-of-life concerns. We will then conduct a randomized trial of a novel HIV Navigation Program, which will be a modification of an existing navigation program that uses trained and experienced volunteers as a core component, offered by a large, comprehensive hospice and palliative care organization. The specific aims of this study are 1) to identify needs and preferences for palliative care and advance care planning of PLWHA, in order to tailor an existing Patient Navigation Program to the specific needs of PLWHA with chronic conditions; and 2) to test the effect of an HIV Patient Navigation Program intervention on outcomes of quality of life, symptom burden, coping ability, and advance care planning; and 3) to determine if effectiveness of the HIV Navigation Program intervention differs by age, gender, ethnicity, education, income level, and level of palliative care service need. Because of the increasing prevalence of HIV coexisting with chronic conditions, there is an urgent need to assess palliative care needs and preferences of PLWHA and design effective interventions. This interdisciplinary study will test, at the community level, a novel health service designed to meet the unique needs of chronically ill PLWHA, and improve and support advance care planning. Results from this study will increase understanding of who are PLWHA at highest risk for need of palliative services and provide a model for providing early palliative care support for PLWHA.

ELIGIBILITY:
Inclusion Criteria:

* HIV dx for 2+ years
* English speaking
* lives within 50 miles of study headquarters
* at least one physical co-morbid condition
* receiving primary care at Institutional Review Board (IRB) approved clinic recruitment site

Exclusion Criteria:

* currently enrolled in hospice care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2013-06; Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Quality of Life | Participants will be followed for 36 months, with quality of life measured at baseline and change from baseline at 9mo, 18mo, 27mo, 36mo
  Using HIV/AIDS Targeted Quality of Life (HAT_QoL) Instrument. It has 34 items measuring 9 dimensions of quality of life on a continuous scale of 0 (worst) to 10 (best).
Symptom burden | Participants will be followed for 36 months with symptom burden measured at baseline and change from baseline at 9mo, 18mo, 27mo, 36mo
  Symptom burden (type and intensity of symptoms) using the Edmonton Symptom Assessment Scale, which has 10 items to measure a total of 10 symptoms on a continuous scale of 0 (no symptom present) to 10 (most severe level).
Coping ability | Participants will be followed for 36 months with coping ability measured at baseline and change from baseline at 9mo, 18mo, 27mo, 36mo
  The Brief COPE will be used to measure illness coping ability. It measures 14 different coping constructs on a scale of 1 (I haven't been doing this at all) to 4 (I've been doing this a lot).
Advance Care Planning | Participants will be assessed at baseline and up to every 6 months over a 36-month period for evidence of completion of advance care planning (yes/no)
  Advance care planning evidenced by number of participants completing an advance directive (living will and/or health proxy/health care power of attorney), or other documentation of initiation and/or implementation of advance care planning.

CONTACTS AND LOCATIONS:
Overall Officials: Jacquelyn Slomka, PhD RN, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
A goal of this project is to test a novel health service model that could be replicated in other sites and with other hospice organizations. Therefore, we will share results with HIV clinicians and researchers, and palliative care and hospice clinicians and researchers. For clinical audiences, we will to target national meetings, including the American Academy of Hospice and Palliative Medicine and Hospice and Palliative Nurses Association annual symposium. The National Hospice and Palliative Care Organization is another avenue for dissemination of this model of care. We also expect to use the Center for AIDS Research, where several of the study team members participate, as an opportunity for reaching researchers. Because previous research shows that specific palliative care needs vary among populations, we will make the de-identified data available so that other centers can evaluate similarities and differences from our population in order to apply our findings.

REFERENCES:
- [Background] Centers for Disease Control and Prevention. HIV/AIDS Surveillance Report. US Department of Health and Human Services, Centers for Disease Control and Prevention, 2007, 2009.
- [Background] Merlin JS, Cen L, Praestgaard A, Turner M, Obando A, Alpert C, Woolston S, Casarett D, Kostman J, Gross R, Frank I. Pain and physical and psychological symptoms in ambulatory HIV patients in the current treatment era. J Pain Symptom Manage. 2012 Mar;43(3):638-45. doi: 10.1016/j.jpainsymman.2011.04.019. Epub 2011 Nov 23. PMID 22115794
- [Background] Fausto JA Jr, Selwyn PA. Palliative care in the management of advanced HIV/AIDS. Prim Care. 2011 Jun;38(2):311-26, ix. doi: 10.1016/j.pop.2011.03.010. PMID 21628041
- [Background] Karus D, Raveis VH, Alexander C, Hanna B, Selwyn P, Marconi K, Higginson I. Patient reports of symptoms and their treatment at three palliative care projects servicing individuals with HIV/AIDS. J Pain Symptom Manage. 2005 Nov;30(5):408-17. doi: 10.1016/j.jpainsymman.2005.04.011. PMID 16310615